CLINICAL TRIAL: NCT03706625
Title: Integrated Discovery of New Immuno-Molecular Actionable Biomarkers for Tumors With Immune-suppressed Environment
Acronym: IDeATIon
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI18022J; 2018-A01099-46 (Other: IDRCB)
Record Dates: First submitted 2018-08-10; First posted 2018-10-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Non Hodgkin Lymphoma; Non Small Cell Lung Cancer; Glioma
Keywords: Non Hodgkin Lymphoma; glioma; lung cancer; HIV; transplantation; brain
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Carcinoma, Non-Small-Cell Lung; Glioma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva, biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Non-Hodgkin-Lymphoma (after transplantation): Immune-suppressed patients suffering from Non-Hodgkin-Lymphoma (after transplantation) and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA)
- Non-small cell lung cancer: Immune-suppressed patients suffering from HIV-related non-small cell lung cancer, followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA)
- Primary Central Nervous System Lymphoma: Patients suffering from primitive cerebral lymphomas and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA)
- Gliomas: Patients suffering from Gliomas and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA)
- Non-Hodgkin-Lymphoma with HIV infection: Immune-suppressed patients (during HIV infection) and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA)
- Immunocompetent Non-Hodgkin-Lymphoma: Immunocompetent patients and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA).
- Immunocompetent Non-small cell lung cancer: Immunocompetent patients suffering from non-small cell lung cancer and followed in the four centers of reference for rare cancers (KVirogref, CANCERVIH, LOC and POLA).

SUMMARY:
The explosion of novel therapies targeting tumor mutations or immune molecules requests to define or better characterize the mutational profiles of tumors that are none or insufficiently explored so far. This is particularly the case for tumors arising in immune-suppressed individuals or environments which have been poorly, if any, analyzed so far with modern molecular methods. The goal of the translational research program, Ideation, is to define novel biomarkers such as the tumor mutational profiling and immunomutanome in such contexts and to compare the results obtained to those observed in immune competent individuals. In addition, this approach will allow to characterize novel key non-invasive diagnostic and prognostic biomarkers such as circulating tumoral DNA and cells. Altogether results will provide novel biomarkers to better adapt therapeutic strategies in these cancers, to monitor response to treatment as well as to define new molecular targets of potential therapeutic strategies.

DETAILED DESCRIPTION:
The main objective is to discover novel invasive and non-invasive immuno-molecular actionable biomarkers in rare but severe tumors arising in immune-suppressed compared for some tumors in immune-competent patients. Indeed, this tumors present a deficient immune environment, either due to the host acquired immune deficiency, i.e. transplantations or HIV infection, or because the diseased tissue belongs in an immune sanctuary as the brain. The primary hypothesis, in this context, is that these tumor mutational profiles and their changes during drug therapy must be influenced by the immune environment and response. This must lead to differences from similar tumors observed in immune-competent environments (immunocompetent individuals or tissues expressing immunity), responsible for: modification in the molecular targets for appropriate drugs ; alteration of tumor immunogenicity and of future immune-based therapies ; specific biomarkers for monitoring the response to drug therapy. The objectives of this program are to carry on invasive and non-invasive investigations in order to define the mutational profile of these free types of severe tumors, non-Hodgkin lymphoma (NHL), lung cancers and gliomas arising in hosts or tissues with altered immunity. These investigations will lead to : identify novel invasive and non-invasive biomarkers for predicting and evaluating efficacy of future personalized and immune-based therapies; compare tumors from immune-suppressed and immune-competent hosts; discover hot spots of tumoral mutations as mechanisms of tumors resistance, new molecular targets for future molecular and immune-bases therapeutic strategies; define the tumor immunomutanome as a score of neo-epitopes predicting: tumor immunogenicity, disease outcome and efficacy of immunotherapies; detect non-invasive tumoral biomarkers from liquid biopsies based on Circulating tumoral DNA and Circulating tumoral Cells to facilitate future diagnosis and monitoring of such tumors; identify biomarkers of tumor escape or resistance to treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Followed at Pitié-Salpêtrière hospital, Tenon hospital, Henri Mondor hospital, Saint-Louis hospital or intercommunal hospital center of Créteil
* Histological diagnosis confirmed of:

  * Non-small cell lung cancer (adenocarcinoma, squamous cell, large cells) related to HIV, or
  * Immunocompetent non-small cell lung cancer (adenocarcinoma, squamous cell, large cells), or
  * Non-Hodgkin's lymphoma (NHL): HIV-related NHL, post-transplant lymphoproliferation (LPT) according to WHO (World Health Organization) 2016 classification, primary CNS (central nervous system) lymphoma (LPS), or
  * Primary CNS lymphoma
  * Immunocompetent NHL: diffuse large B cell lymphoma (ABC or GC)
  * Glioma
* Naïve cancer treatment (except for the specific case of gliomas with certain or possible activation of MAPK (Mitogen-activated protein kinases) and MMR (Mismatch Repair) inactivation).
* Cancer undergoing surgery for excision or a large biopsy (pleural biopsy under video-thoracoscopy, mediastinoscopy, biopsy lymph node excision or cutaneous or cerebral metastasis).
* For patients with NSCLC: hemoglobin level> 9 g / dL; for patients with NHL or glioma: hemoglobin > 7 g / dL.
* Weight ≥ 48 kg.
* Informed consent to participation signed before carrying out any specific procedure of the study.
* Affiliation to the French social security system.

Exclusion Criteria:

* Other cancer than those in the study:

  * For NHL after transplantation: marginal zone NHL, follicular NHL, mantle cell NHL, lymphoplasmocytic NHL (non-WHO lymphoma as LPT)
  * For HIV-related LPTs and NHLs: LPS
  * For LPT: tumor EBV status unknown
  * For immunocompetent NHL: other NHL than diffuse large B cell lymphoma
  * For lung cancers: small cell lung cancer
* Absence of tumor material, blood or saliva samples taken before the start of chemotherapy (except for the specific case of gliomas with certain or possible activation of MAPK and MMR inactivation)
* Major under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed-up at Pitié-Salpêtrière hospital, Tenon hospital, Henri Mondor hospital, Saint-Louis hospital or intercommunal hospital center of Créteil with histological diagnosis of HIV-related non-small cell lung cancer, immunocompetent non-small cell lung cancer, HIV-related Non-Hodgkin-Lymphomas (NHL), immunocompetent NHL, post-transplant NHL, primary lymphoma of the central nervous system, glioma.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the tumor invasive biomarkers | at Day 0
  Analyze of the tumor biomarkers on frozen biopsy for the three types of cancer (NHL, lung cancer and glioma)

SECONDARY OUTCOMES:
Determination of tumoral biomarkers | at Day 0
  i) the mutational tumor profile by using a next generation sequencing (NGS) comparingson of the tumor DNAgenome with the patient's constitutional genome (sequenced on blood or saliva) for the three types of cancer (NHL, lung cancer and glioma) and ii) immunomutanome and score of neo-epitopes defined by tumor RNA-sequencing defining the specific mutants expressed in the tumor and able to be recognized by the immune system.
Prognostic value of the tumor non invasive biomarkers | at Day 0, Month 3 and Month 6
  The analysis of circulating DNA (ctDNA) will be performed from plasma collected from the prospective cohort of the patients for the three types of cancer (NHL, lung cancer and glioma). DNA will be extracted and amplified followed by Next-Generation Sequencing (NGS) and Droplet digital PCR (ddPCR) analysis for the identification of new biomarkers and/or for the follow up of mutations previously identified on tumor DNA. Results will be compared to tissue results in each group and to CTCs results in the Lung cancer group and prognostic values of these biomarkers will be assessed from clinical datas.
Prognostic value of the tumor non-invasive biomarkers | at Day 0, Month 3 and Month 6
  The analysis of circulating tumor cells (CTCs) will be performed from whole peripheral blood collected from the prospective cohort of patients with lung cancer infected or not with HIV. CTC fraction will be prepared from a cell size-based enrichment protocol. Then, DNA and RNA will be extracted and amplified followed by Next-Generation Sequencing (NGS) and RNA sequencing for the identification of new biomarkers. Droplet digital PCR (ddPCR) analysis will also be performed for validation and patient follow-up. Mutations and expression data in CTC will be compared to tissue and ctDNA in the two groups and prognostic values of these biomarkers will be assessed from clinical datas.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe SPANO, MD, PhD, Study Chair — Pitié-Salpêtrière hospital (APHP)
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.